CLINICAL TRIAL: NCT05644054
Title: The Impact of THC on Pain Modulation in Fibromyalgia: A Cross-Over, Randomized, Double-Blind Placebo-Controlled Study
Brief Title: The Impact of THC on Pain Modulation in Fibromyalgia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv Medical Center (Other)
Responsible Party: Principal Investigator, yara agbaria, researcher, Tel Aviv Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TLV-16-320
Record Dates: First submitted 2022-11-21; First posted 2022-12-09 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Fibromyalgia, Primary
MeSH Terms: conditions — Fibromyalgia | interventions — Dronabinol

STUDY DESIGN:
Intervention Model Description: A Cross-Over, Double-Blind Placebo-Controlled Study
Who Masked: Participant, Investigator
Masking Description: Neither the participants nor the investigators will be aware of the drug being administered.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (THC) - session 1 (Experimental): Patients will attend two sessions in a crossover design, where they will receive one of the drugs in a randomized sequence at each session.
  Interventions: Drug: THC
- Placebo - session 2 (Placebo Comparator): Patients will attend two sessions in a crossover design, where they will receive one of the drugs in a randomized sequence at each session.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THC — Patients will be administered a one-time dosage of 0.2 mg/kg THC oil (AXIBAN, T10/C2, manufactured by Panaxia Pharmaceuticals, Lod, Israel)
  Arms: Treatment (THC) - session 1
Drug: Placebo — Patients will be administered a one-time dosage of 0.2 mg/kg of a placebo consisting of an inactive oil.
  Arms: Placebo - session 2

SUMMARY:
The objective of this cross-sectional, double-blind, placebo-controlled clinical trial is to enhance our understanding of the pain modulation mechanisms in females diagnosed with Fibromyalgia syndrome (FMS).

This study is designed to address several key questions:

1. Is there a discernible difference in the effectiveness of the two prevalent pain modulation approaches, namely Conditioned Pain Modulation (CPM) and Offset Analgesia (OA), in individuals with FMS? To answer this, both FMS patients and an age- and sex-matched healthy control group will engage in these paradigms outside of the MRI scanner.
2. How does Tetrahydrocannabinol (THC) influence CPM and OA in FMS patients? Here, the study will observe the performance of FMS patients in both paradigms after receiving treatments with THC and a placebo, conducted outside the scanner.
3. What neural alterations in pain modulation circuits are triggered by THC? To investigate this, FMS patients will undergo the OA test inside the MRI scanner following both THC and placebo treatments.
4. How does THC affect resting-state brain function in FMS patients? This part of the study involves resting-state brain scans to measure changes in functional connectivity following treatments with THC and a placebo.

DETAILED DESCRIPTION:
Fibromyalgia syndrome (FMS) is a condition marked by pervasive chronic pain throughout the musculoskeletal system, often accompanied by chronic sleep disturbances, fatigue, memory challenges, and more. Despite significant advancements in the understanding of pain mechanisms due to breakthroughs in neuroscience and pain medicine, current treatments for FMS fall short of providing adequate relief, leaving many patients battling ongoing pain and related symptoms.

The complete pathophysiology of FMS remains elusive, but there is substantial evidence indicating the involvement of various factors, including central sensitization and impaired descending pain modulation pathways as evidenced by functional imaging studies and sensory tests such as conditioned pain modulation (CPM) and offset analgesia (OA). Given this, comprehending the pathophysiology of FMS and the mechanisms involved is crucial. Additionally, it is critical to understand how new treatments can influence pain modulation in FMS.

Recent research increasingly supports the use of cannabis, particularly Tetrahydrocannabinol (THC), for alleviating chronic pain in various syndromes. Yet, there's a lack of extensive research exploring its effectiveness in randomized, double-blind trials. Exploring THC's effects in clinical pain models could enhance our understanding of pain regulation in FMS.

The current study aims to deepen our understanding of sensory and neural mechanisms in FMS, employing quantitative sensory testing such as CPM and OA, and fMRI. A key objective is to ascertain the impact of THC on pain modulation in FMS within a double-blind controlled framework.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with fibromyalgia for over 3 months according to American college of rheumatology
2. Do not respond well to analgesic medications and or have severe side effects
3. Medium to high level of pain (over 40 on visual analogue scale scale)
4. Does not have other pain-related syndromes
5. Not treated regularly with cannabis.
6. Is ready to stop taking central nervous system medications 3 days prior to the experiment.

Exclusion Criteria:

1. alleviated levels of anxiety (above 52 in STAI)
2. Psychiatric medications due to psychiatric diagnoses (depression, bi-polar syndrome, etc.).
3. Cardiovascular problems
4. Neurological diseases (other than migraine).
5. Pregnancy or breastfeeding
6. Alcoholism or substance abuse
7. Cancer
8. Blood pressure problems
9. Patients that used cannabis in the past month
10. Illegibility to MRI

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 40 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Functional Connectivity (FC) | 2 hours after drug administration
  The variations in FC measured during the resting-state scan will be assessed using within-between network connectivity at baseline and following treatments with either THC or a placebo in FMS patients.
Blood Oxygenation Level (BOLD) | 2 hours after drug administration
  The variations in BOLD activity measured during the sensory test will be assessed using ROI to ROI analysis at baseline and following treatments with either THC or a placebo in FMS patients.
Quantitative Sensory Tests: Conditioned pain modulation (CPM) and offset analgesia (OA) magnitude | 2 hours after drug administration
  Baseline assessments of CPM and OA magnitude will be conducted for both FMS patients and their corresponding healthy control group. Furthermore, the magnitude of these tests will also be evaluated after administering either THC or placebo treatments in FMS patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Ablin, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No